CLINICAL TRIAL: NCT04180527
Title: Reducing Patient Anxiety Through Patients Telling Their Stories
Brief Title: Preoperative Hip Knee Anxiety Sleep Study
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Gary E. Loyd, Senior Staff Anesthesiologist; Director of Perioperative Surgical Home, Henry Ford Health System
Other Study IDs: 12849
Record Dates: First submitted 2019-11-20; First posted 2019-11-27 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Anxiety; Sleep; Surgery
Keywords: preoperative; sleep; anxiety; hip surgery; knee surgery; storytelling
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Quality Improvement Initiative: This group of patients have not received previous patients' stories about their hip or knee surgery before undergoing their own hip or knee surgery.
- Post-Quality Improvement Initiative: This group of patients have received previous patients' stories regarding about their hip or knee surgery before undergoing their own hip or knee surgery.

SUMMARY:
This study is about assessing the impact of reading previous patients' stories related to their hip or knee replacement surgery on patients' preoperative anxiety and sleep. This provision of previous patients' stories is part of an ongoing perioperative QI project in the regional anesthesiology division.

DETAILED DESCRIPTION:
This will be a pre-post experimental design study. The pre-intervention group of 80 hip or knee replacement surgery patients will receive the Amsterdam Preoperative Anxiety and Information Scale (APAIS) and Pittsburgh Sleep Quality Index (PSQI) in Preop Holding prior to having their block for their surgery. The block resident will give and collect the scale and inventory to patients. Patients are given these surveys as part of a quality improvement initiative, independently of this study. The survey data will be entered into the secure electronic research database. Following this, the post-intervention group of 80 patients will be given copies of previous patients' stories at their last visit to the surgeon's office prior to their surgery. These stories will be administered to all hip and knee surgery patients as part of the new standard of care due to a perioperative QI initiative, independently of this study taking place. These subjects will also receive the APAIS and PSQI for assessment in Preop Holding prior to their block for surgery, as part of the new standard of care. A third party broker will then de-identify the survey data and provide it to the research team for analysis. A two-sided independent t-test will be performed to evaluate the differences in anxiety and sleep scores between the pre- and post-intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Planned to undergo a hip or knee replacement surgery at Henry Ford Hospital

Exclusion Criteria:

* Diagnoses involving sleep disturbance or psychiatric anxiety

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will focus on patients who undergo full hip or knee arthroplasty at Henry Ford Hospital and do not have any diagnoses involving sleep disturbance or psychiatric anxiety.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Determine the impact of story reading on preoperative anxiety in hip and knee surgery patients | 15 minutes
  Compare preoperative Amsterdam Preoperative Anxiety and Information Scale (APAIS) scores of patients undergoing hip or knee surgery who have read previous patients' stories to those who have not read the stories. The APAIS anxiety anxiety scale can have a range from 4 to 20, with higher scores indicating a higher anxiety score. The cutoff score for identifying anxious patients in a clinical practice is typically 11.
Determine the impact of story reading on preoperative sleep in hip and knee surgery patients | 15 minutes
  Compare preoperative Pittsburgh Sleep Quality Index scores of patients undergoing hip or knee surgery who have read previous patients' stories to those who have not read the stories.The PSQI score can range from a minimum of 0 and a maximum of 21, with a score of 5 or higher being indicative of poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771